CLINICAL TRIAL: NCT04874415
Title: Behavioral Economics for Activity Motivation in Adolescents and Young Adults With Prediabetes and Type 2 Diabetes
Brief Title: Behavioral Economics for Activity Motivation in Adolescents (BEAM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mary Ellen Vajravelu, MD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: STUDY21040122; K23DK125719-01 (NIH)
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes; PreDiabetes; Insulin Resistance; Polycystic Ovary Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Insulin Resistance; Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): 1RLD=One text per day, ramped goal, loss incentive, daily goal time period.
  Interventions: Behavioral: 1RLD
- Condition 2 (Experimental): 1RLW=One text per day, ramped goal, loss incentive, weekly goal time period.
  Interventions: Behavioral: 1RLW
- Condition 3 (Experimental): 1RGD=One text per day, ramped goal, gain incentive, daily goal time period.
  Interventions: Behavioral: 1RGD
- Condition 4 (Experimental): 1RGW=One text per day, ramped goal, gain incentive, weekly goal time period.
  Interventions: Behavioral: 1RGW
- Condition 5 (Experimental): 2RLD=Two texts per day, ramped goal, loss incentive, daily goal time period.
  Interventions: Behavioral: 2RLD
- Condition 6 (Experimental): 2RLW=Two texts per day, ramped goal, loss incentive, weekly goal time period.
  Interventions: Behavioral: 2RLW
- Condition 7 (Experimental): 2RGD=Two texts per day, ramped goal, gain incentive, daily goal time period.
  Interventions: Behavioral: 2RGD
- Condition 8 (Experimental): 2RGW=Two texts per day, ramped goal, gain incentive, weekly goal time period.
  Interventions: Behavioral: 2RGW
- Condition 9 (Experimental): 1FLD=One text per day, fixed goal, loss incentive, daily goal time period.
  Interventions: Behavioral: 1FLD
- Condition 10 (Experimental): 1FLW=One text per day, fixed goal, loss incentive, weekly goal time period.
  Interventions: Behavioral: 1FLW
- Condition 11 (Experimental): 1FGD=One text per day, fixed goal, gain incentive, daily goal time period.
  Interventions: Behavioral: 1FGD
- Condition 12 (Experimental): 1FGW=One text per day, fixed goal, gain incentive, weekly goal time period.
  Interventions: Behavioral: 1FGW
- Condition 13 (Experimental): 2FLD=Two texts per day, fixed goal, loss incentive, daily goal time period.
  Interventions: Behavioral: 2FLD
- Condition 14 (Experimental): 2FLW=Two texts per day, fixed goal, loss incentive, weekly goal time period.
  Interventions: Behavioral: 2FLW
- Condition 15 (Experimental): 2FGD=Two texts per day, fixed goal, gain incentive, daily goal time period.
  Interventions: Behavioral: 2FGD
- Condition 16 (Experimental): 2FGW=Two texts per day, fixed goal, gain incentive, weekly goal time period.
  Interventions: Behavioral: 2FGW

INTERVENTIONS:
Behavioral: 1RLD — 1RLD=One text per day, ramped goal, loss incentive, daily goal time period
  Arms: Condition 1
Behavioral: 1RLW — 1RLW=One text per day, ramped goal, loss incentive, weekly goal time period.
  Arms: Condition 2
Behavioral: 1RGD — 1RGD=One text per day, ramped goal, gain incentive, daily goal time period.
  Arms: Condition 3
Behavioral: 1RGW — One text per day, ramped goal, gain incentive, weekly goal time period.
  Arms: Condition 4
Behavioral: 2RLD — Two texts per day, ramped goal, loss incentive, daily goal time period.
  Arms: Condition 5
Behavioral: 2RLW — Two texts per day, ramped goal, loss incentive, weekly goal time period.
  Arms: Condition 6
Behavioral: 2RGD — Two texts per day, ramped goal, gain incentive, daily goal time period.
  Arms: Condition 7
Behavioral: 2RGW — Two texts per day, ramped goal, gain incentive, weekly goal time period.
  Arms: Condition 8
Behavioral: 1FLD — One text per day, fixed goal, loss incentive, daily weekly goal time period.
  Arms: Condition 9
Behavioral: 1FLW — One text per day, fixed goal, loss incentive, weekly goal time period.
  Arms: Condition 10
Behavioral: 1FGD — One text per day, fixed goal, gain incentive, daily goal time period.
  Arms: Condition 11
Behavioral: 1FGW — One text per day, fixed goal, gain incentive, weekly goal time period.
  Arms: Condition 12
Behavioral: 2FLD — Two texts per day, fixed goal, loss incentive, daily goal time period.
  Arms: Condition 13
Behavioral: 2FLW — Two texts per day, fixed goal, loss incentive, weekly goal time period.
  Arms: Condition 14
Behavioral: 2FGD — Two texts per day, fixed goal, gain incentive, daily goal time period.
  Arms: Condition 15
Behavioral: 2FGW — Two texts per day, fixed goal, gain incentive, weekly goal time period.
  Arms: Condition 16

SUMMARY:
There is an urgent need to engineer targeted physical activity interventions that are effective and scalable for obese adolescents and young adults (AYA) with type 2 diabetes (T2D), who often have very low levels of physical activity. The BEAM Trial is a mobile health (mHealth) intervention that uses behavioral economic-informed financial incentives and text messaging to promote physical activity in AYA with T2D and prediabetes.

DETAILED DESCRIPTION:
Some secondary outcome measures from the protocol were inadvertently left out when creating the registration and have been added with the results.

ELIGIBILITY:
Inclusion Criteria:

* 1) Males or females age 13 to 22 years.
* 2) Overweight or obese (BMI ≥85th percentile for age/sex, or ≥25 kg/m2 for participants ≥18 years)
* 3) Diagnosis with prediabetes or type 2 diabetes
* 4) Consent (subjects 18 and older), Parental/guardian permission (subjects 13-17), assent (subjects 13-17)
* 5) Willingness to wear Fitbit during waking hours daily for duration of run-in and intervention.
* 6) Possession of a smartphone.

Exclusion Criteria:

* 1) Potential subject unable to speak or read in English
* 2) Severe cognitive impairment
* 3) Permanent or temporary physical disability that impairs ambulation or precludes engagement in MVPA
* 4) Current pregnancy
* 5) Previously-diagnosed or current restrictive or purging eating disorder
* 6) Moderate to vigorous physical activity (MVPA) >30 minutes per day or Fitbit wear < 4 days during second week of 2-week run-in period

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: n=75 participants signed consent to participate in the study. n=74 completed the baseline study visit and 2-week run-in using Fitbit. Those with insufficient Fitbit data or more than 30 minutes of moderate-vigorous physical activity daily were excluded prior to randomization (n=7).
Groups:
- 1RLD: One text per day, ramped goal, loss incentive, daily goal time period
- 1RLW: One text per day, ramped goal, loss incentive, weekly goal time period.
- 1RGD: One text per day, ramped goal, gain incentive, daily goal time period.
Period: Overall Study
Arm/Group | 1FLD | 1FLW | 1RLD | 1RLW | 1FGD | 1FGW | 1RGD | 1RGW | 2FLD | 2FLW | 2RLD | 2RLW | 2FGD | 2FGW | 2RGD | 2RGW
Started | 5 | 4 | 4 | 5 | 4 | 3 | 3 | 4 | 4 | 5 | 5 | 4 | 4 | 4 | 5 | 4
Completed | 3 | 3 | 3 | 3 | 2 | 2 | 2 | 2 | 0 | 2 | 3 | 3 | 3 | 3 | 1 | 3
Not Completed | 2 | 1 | 1 | 2 | 2 | 1 | 1 | 2 | 4 | 3 | 2 | 1 | 1 | 1 | 4 | 1
Not completed — Missing Fitbit data but not lost to follow up | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 1 | 4 | 0
Not completed — Missing Fitbit data and lost to follow up | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 1
Not completed — Did not attend final study visit but had Fitbit data | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1FLD | 1FLW | 1RLD | 1RLW | 1FGD | 1FGW | 1RGD | 1RGW | 2FLD | 2FLW | 2RLD | 2RLW | 2FGD | 2FGW | 2RGD | 2RGW | Total
Number analyzed (Participants) | 5 | 4 | 4 | 5 | 4 | 3 | 3 | 4 | 4 | 5 | 5 | 4 | 4 | 4 | 5 | 4 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.1 (1.8) | 15.2 (2.6) | 15.3 (1.0) | 15.0 (1.3) | 15.9 (1.6) | 15.2 (1.9) | 16.7 (3.3) | 17.0 (2.7) | 17.5 (2.5) | 16.3 (1.0) | 17.7 (2.0) | 17.2 (3.2) | 16.0 (0.6) | 14.1 (0.9) | 16.1 (1.3) | 15.8 (2.5) | 16.1 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 4 | 2 | 1 | 3 | 2 | 3 | 2 | 2 | 2 | 3 | 2 | 4 | 3 | 45
  Male | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 1 | 3 | 3 | 2 | 1 | 2 | 1 | 1 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Non-Hispanic Black | 2 | 2 | 1 | 3 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 2 | 3 | 0 | 22
  Non-Hispanic Native American/Alaskan Native/Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Non-Hispanic White | 1 | 0 | 2 | 2 | 2 | 2 | 1 | 2 | 1 | 3 | 2 | 3 | 3 | 2 | 2 | 3 | 31
  Hispanic/Latino/Latina | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Multiracial | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 9
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 38.4 [35.4 to 48.0] | 43.6 [41.9 to 50.3] | 43.7 [36.6 to 46.6] | 34.9 [34.7 to 35.6] | 46.9 [42.4 to 52.9] | 38.3 [36.3 to 42.3] | 40.3 [31.6 to 41.7] | 42.1 [35.2 to 45.4] | 39.6 [37.7 to 44.0] | 34.7 [32.8 to 36.8] | 44.6 [40.6 to 45] | 40.2 [34.1 to 48] | 37.8 [35.8 to 45.8] | 35.5 [31.6 to 39.5] | 35.9 [33 to 41.1] | 34.5 [28.9 to 44.2] | 40 [34.7 to 44.6]

OUTCOME MEASURES:

1. Primary Outcome: Change in Moderate to Vigorous Physical Activity (MVPA)
Description: Effects of time spent in MVPA was measured by assessing the change in weekly mean minutes in MVPA per day from baseline
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per day
Groups:
- Once Daily Text Message: All participants assigned to once (versus twice) daily text messages, including 1FLD, 1FLW, 1RLD, 1RLW, 1FGD, 1FGW, 1RGD, 1RGW.
- Twice Daily Text Message: All participants assigned to twice (versus once) daily text messages, including 2FLD, 2FLW, 2RLD, 2RLW, 2FGD, 2FGW, 2RGD, 2RGW.
- Fixed Step Count Goal: All participants assigned to fixed (versus ramped) step count goal, including 1FLD, 1FLW, 1FGD, 1FGW, 2FLD, 2FLW, 2FGD, 2FGW,
- Ramped Step Count Goal: All participants assigned to ramped (versus fixed) step count goal, including 1RLD, 1RLW, 1RGD, 1RGW, 2RLD, 2RLW, 2RGD, 2RGW,
- Loss Framed Incentive: All participants assigned to loss (versus gain) framed incentive, including 1FLD, 1FLW, 1RLD, 1RLW, 2FLD, 2FLW, 2RLD, 2RLW
- Gain Framed Incentive: All participants assigned to gain (versus loss) framed incentive, including 1FGD, 1FGW, 1RGD, 1RGW, 2FGD, 2FGW, 2RGD, 2RGW
- Daily Step Count Goal: All participants assigned to daily (versus weekly) step count goal, including 1FLD, 1FGD, 1RLD, 1RGD, 2FLD, 2FGD, 2RLD, 2RGD
- Weekly Step Count Goal: All participants assigned to weekly (versus daily) step count goal, including 1FLW, 1FGW, 1RLW, 1RGW, 2FLW, 2FGW, 2RLW, 2RGW
Arm/Group | Once Daily Text Message | Twice Daily Text Message | Fixed Step Count Goal | Ramped Step Count Goal | Loss Framed Incentive | Gain Framed Incentive | Daily Step Count Goal | Weekly Step Count Goal
Number analyzed (Participants) | 21 | 18 | 19 | 20 | 20 | 19 | 18 | 21
minutes per day
  Baseline | 6.1 [3.6 to 8.6] | 7.1 [3.0 to 11.3] | 5.0 [1.8 to 8.2] | 8.2 [3.7 to 12.8] | 5.1 [2.0 to 8.1] | 8.2 [3.6 to 12.7] | 6.5 [3.3 to 9.7] | 6.7 [3.1 to 10.3]
  Change from baseline to 12 weeks | 2.3 [-0.9 to 5.5] | 1.8 [-2.9 to 6.5] | 3.3 [-0.9 to 7.4] | 0.8 [-4.0 to 5.7] | 4.0 [-0.2 to 8.3] | 0.07 [-4.7 to 4.9] | -0.2 [-3.1 to 2.8] | 4.3 [-0.5 to 9.0]
Statistical Analysis 1: Comparison: Once Daily Text Message vs Twice Daily Text Message; Test type: Superiority — Main effects of each intervention factor were estimated using linear regression including all prespecified two-way interactions; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-6.2 to 5.3] — Once daily text message is reference group. Least-squares means (marginal means) were calculated, averaging across levels of the other factors with equal weighting (asbalanced)
Statistical Analysis 2: Comparison: Fixed Step Count Goal vs Ramped Step Count Goal; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-9.4 to 4.6] — Fixed step count is reference group. Least-squares means (marginal means) were calculated, averaging across levels of the other factors with equal weighting (asbalanced)
Statistical Analysis 3: Comparison: Loss Framed Incentive vs Gain Framed Incentive; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-11 to 3.1] — Loss framed incentive is reference group. Least-squares means (marginal means) were calculated, averaging across levels of the other factors with equal weighting (asbalanced)
Statistical Analysis 4: Comparison: Daily Step Count Goal vs Weekly Step Count Goal; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.4, 95% CI 2-sided [-1.0 to 9.8] — Daily step count goal is reference group. Least-squares means (marginal means) were calculated, averaging across levels of the other factors with equal weighting (asbalanced)

2. Secondary Outcome: Change in Daily Step Count
Description: Daily step count will be measured by assessing the change in daily mean steps from baseline
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: steps
Arm/Group | Once Daily Text Message | Twice Daily Text Message | Fixed Step Count Goal | Ramped Step Count Goal | Loss Framed Incentive | Gain Framed Incentive | Daily Step Count Goal | Weekly Step Count Goal
Number analyzed (Participants) | 21 | 18 | 19 | 20 | 20 | 19 | 18 | 21
steps | 962 [-446 to 2369] | 276 [-1486 to 2038] | 1789 [144 to 3433] | -551 [-2201 to 1099] | 1266 [53 to 2478] | -28 [-1852 to 1797] | 687 [-959 to 2332] | 551 [-973 to 2076]
Statistical Analysis 1: Comparison: Once Daily Text Message vs Twice Daily Text Message; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -686, 95% CI 2-sided [-2997 to 1626] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fixed Step Count Goal vs Ramped Step Count Goal; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2340, 95% CI 2-sided [-4794 to 115] — Fixed step count goal is reference group. Least-squares means (marginal means) were calculated, averaging across levels of the other factors with equal weighting (asbalanced)
Statistical Analysis 3: Comparison: Loss Framed Incentive vs Gain Framed Incentive; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1293, 95% CI 2-sided [-3477 to 890]; Loss framed incentive is reference group. Least-squares means (marginal means) were calculated, averaging across levels of the other factors with equal weighting (asbalanced)
Statistical Analysis 4: Comparison: Daily Step Count Goal vs Weekly Step Count Goal; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -135, 95% CI 2-sided [-2424 to 2153] — [estimate comment as in outcome 1, analysis 4]

3. Secondary Outcome: Change in BMI Z-score
Description: Z-score calculated using "zanthro" package in Stata, according to U.S. CDC growth charts. The BMI Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched adolescents and young adults). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population. A Z-score of 0 represents the population mean. BMI Z-scores greater than 1.645 are consistent with pediatric obesity.
Time Frame: From baseline to follow-up in-person study visits, separated by 3 months
Population: Participants were censored if they started weight-altering medications, including glucagon-like peptide-1 receptor agonists, metformin, or insulin (n=4). BMI Z-scores were not calculated for individuals older than 20 years (n=1)
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Once Daily Text Message | Twice Daily Text Message | Fixed Step Count Goal | Ramped Step Count Goal | Loss Framed Incentive | Gain Framed Incentive | Daily Step Count Goal | Weekly Step Count Goal
Number analyzed (Participants) | 26 | 24 | 26 | 24 | 25 | 25 | 26 | 24
Z-score | -0.02 [-0.05 to 0.01] | -0.03 [-0.06 to 0.01] | -0.009 [-0.04 to 0.02] | -0.03 [-0.07 to -0.005] | -0.03 [-0.06 to -0.001] | -0.01 [-0.04 to 0.02] | -0.02 [-0.05 to 0.007] | -0.02 [-0.05 to 0.007]
Statistical Analysis 1: Comparison: Once Daily Text Message vs Twice Daily Text Message; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.05 to 0.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fixed Step Count Goal vs Ramped Step Count Goal; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.07 to 0.02] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Loss Framed Incentive vs Gain Framed Incentive; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.02 to 0.06]; [other analysis details as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Daily Step Count Goal vs Weekly Step Count Goal; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.0006, 95% CI 2-sided [-0.04 to 0.04] — [estimate comment as in outcome 1, analysis 4]

4. Secondary Outcome: Change in Plasma Glucose
Description: mg/dL; obtained fasting
Time Frame: From baseline to follow-up in-person study visits, separated by 3 months
Population: Participants were censored if they started weight-altering medications, including glucagon-like peptide-1 receptor agonists, metformin, or insulin (n=4). Participants who arrived to the second study visit non-fasting had fasting-sensitive laboratory measures censored (n=1). Due to sample processing errors, n=2 additional results were missing.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Once Daily Text Message | Twice Daily Text Message | Fixed Step Count Goal | Ramped Step Count Goal | Loss Framed Incentive | Gain Framed Incentive | Daily Step Count Goal | Weekly Step Count Goal
Number analyzed (Participants) | 25 | 23 | 23 | 25 | 23 | 25 | 25 | 23
mg/dL | 0.006 [-10.3 to 10.3] | 0.000000004 [-0.00001 to 0.00001] | 0.000002 [-0.004 to 0.004] | 0.00001 [-0.03 to 0.03] | 0.000000002 [-0.000007 to 0.000007] | 0.01 [-12.7 to 12.7] | 0.00002 [-0.04 to 0.04] | 0.000001 [-0.003 to 0.003]
Statistical Analysis 1: Comparison: Once Daily Text Message vs Twice Daily Text Message; Test type: Superiority — Main effects were estimated using generalized linear models with log link. No interactions were included (failure to converge); Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-10.3 to 10.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fixed Step Count Goal vs Ramped Step Count Goal; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.00001, 95% CI 2-sided [-0.03 to 0.03] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Loss Framed Incentive vs Gain Framed Incentive; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-12.7 to 12.7] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Daily Step Count Goal vs Weekly Step Count Goal; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.00002, 95% CI 2-sided [-0.03 to 0.03] — [estimate comment as in outcome 1, analysis 4]

5. Secondary Outcome: Change in Insulin
Description: uIU/mL; obtained fasting
Time Frame: From baseline to follow-up in-person study visits, separated by 3 months
Population: Participants were censored if they started weight-altering medications, including glucagon-like peptide-1 receptor agonists, metformin, or insulin (n=4). Due to sample processing errors, n=4 additional results were missing. Participants who arrived to the second study visit non-fasting had fasting-sensitive laboratory measures censored (n=1).
Measure: Least Squares Mean (95% Confidence Interval); unit: uIU/mL
Arm/Group | Once Daily Text Message | Twice Daily Text Message | Fixed Step Count Goal | Ramped Step Count Goal | Loss Framed Incentive | Gain Framed Incentive | Daily Step Count Goal | Weekly Step Count Goal
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 22 | 24 | 23 | 23
uIU/mL | 0.00000002 [-1.5 to 1.5] | 0.00003 [-2313 to 2313] | 0.0000006 [-46 to 46] | 0.000001 [-74 to 74] | 0.005 [-6.8 to 6.9] | 0.0000000001 [-0.02 to 0.02] | 0.3 [-125 to 126] | 0.000000000002 [-0.0003 to 0.0003]
Statistical Analysis 1: Comparison: Once Daily Text Message vs Twice Daily Text Message; Test type: Superiority — Main effects of each intervention factor were estimated using generalized linear models with log link, including all prespecified two-way interactions; Mean Difference (Final Values) = 0.00003, 95% CI 2-sided [-2311 to 2311] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fixed Step Count Goal vs Ramped Step Count Goal; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.0000004, 95% CI 2-sided [-27.9 to 27.9] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Loss Framed Incentive vs Gain Framed Incentive; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-6.9 to 6.8] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Daily Step Count Goal vs Weekly Step Count Goal; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-126 to 125] — [estimate comment as in outcome 1, analysis 4]

6. Secondary Outcome: Change in Hemoglobin A1c
Description: Percent (%)
Time Frame: From baseline to follow-up in-person study visits, separated by 3 months
Population: Participants were censored if they started weight- or glucose-altering medications, including glucagon-like peptide-1 receptor agonists, metformin, or insulin (n=4). Due to sample processing errors, n=2 additional results were missing.
Measure: Least Squares Mean (95% Confidence Interval); unit: % (HbA1c unit)
Arm/Group | Once Daily Text Message | Twice Daily Text Message | Fixed Step Count Goal | Ramped Step Count Goal | Loss Framed Incentive | Gain Framed Incentive | Daily Step Count Goal | Weekly Step Count Goal
Number analyzed (Participants) | 25 | 24 | 25 | 24 | 24 | 25 | 25 | 24
% (HbA1c unit) | 0.003 [-3.9 to 3.9] | 0.00000002 [-0.00007 to 0.00007] | 0.00000003 [-0.0001 to 0.0001] | 0.002 [-2.6 to 2.6] | 0.00001 [-0.03 to 0.03] | 0.000004 [-0.009 to 0.009] | 0.02 [-22.8 to 22.8] | 0.000000002 [-0.000009 to 0.000009]
Statistical Analysis 1: Comparison: Once Daily Text Message vs Twice Daily Text Message; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-3.9 to 3.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fixed Step Count Goal vs Ramped Step Count Goal; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-2.6 to 2.6] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Loss Framed Incentive vs Gain Framed Incentive; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.00001, 95% CI 2-sided [-0.02 to 0.02] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Daily Step Count Goal vs Weekly Step Count Goal; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-22.8 to 22.8] — [estimate comment as in outcome 1, analysis 4]

7. Secondary Outcome: Change in Triglycerides
Description: mg/dL; obtained fasting
Time Frame: From baseline to follow-up in-person study visits, separated by 3 months
Population: Participants were censored if they started weight-altering medications, including glucagon-like peptide-1 receptor agonists, metformin, or insulin (n=4). Due to sample processing errors, n=2 additional results were missing. Participants who arrived to the second study visit non-fasting had fasting-sensitive laboratory measures censored (n=1).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Once Daily Text Message | Twice Daily Text Message | Fixed Step Count Goal | Ramped Step Count Goal | Loss Framed Incentive | Gain Framed Incentive | Daily Step Count Goal | Weekly Step Count Goal
Number analyzed (Participants) | 26 | 22 | 24 | 24 | 24 | 24 | 25 | 23
mg/dL | 0.03 [-38.2 to 38.3] | 0.00000005 [-0.0001 to 0.0001] | 0.00001 [-0.04 to 0.04] | 0.0001 [-0.3 to 0.3] | 0.0006 [-0.8 to 0.8] | 0.000002 [-0.006 to 0.006] | 0.0001 [-0.3 to 0.3] | 0.00001 [-0.04 to 0.04]
Statistical Analysis 1: Comparison: Once Daily Text Message vs Twice Daily Text Message; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-38.3 to 38.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fixed Step Count Goal vs Ramped Step Count Goal; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.0001, 95% CI 2-sided [-0.3 to 0.3] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Loss Framed Incentive vs Gain Framed Incentive; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.0006, 95% CI 2-sided [-0.8 to 0.8] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Daily Step Count Goal vs Weekly Step Count Goal; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.0001, 95% CI 2-sided [-0.4 to 0.4] — [estimate comment as in outcome 1, analysis 4]

8. Secondary Outcome: Change in Low-density Lipoprotein (LDL)
Description: mg/dL; obtained fasting
Time Frame: From baseline to follow-up in-person study visits, separated by 3 months
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Once Daily Text Message | Twice Daily Text Message | Fixed Step Count Goal | Ramped Step Count Goal | Loss Framed Incentive | Gain Framed Incentive | Daily Step Count Goal | Weekly Step Count Goal
Number analyzed (Participants) | 26 | 22 | 24 | 24 | 24 | 24 | 25 | 23
mg/dL | 0.1 [-65.6 to 65.9] | 0.2 [-97.1 to 97.5] | 0.1 [-60.7 to 60.9] | 0.2 [-105 to 105] | 0.005 [-4.6 to 4.6] | 5.7 [-1.3 to 12.8] | 5.4 [-0.7 to 11.6] | 0.005 [-4.9 to 4.9]
Statistical Analysis 1: Comparison: Once Daily Text Message vs Twice Daily Text Message; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-31.4 to 31.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fixed Step Count Goal vs Ramped Step Count Goal; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-44.3 to 44.5] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Loss Framed Incentive vs Gain Framed Incentive; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [-2.7 to 14.2] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Daily Step Count Goal vs Weekly Step Count Goal; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-13.3 to 2.4] — [estimate comment as in outcome 1, analysis 4]

9. Secondary Outcome: Change in High-density Lipoprotein (HDL)
Description: mg/dL; obtained fasting
Time Frame: From baseline to follow-up in-person study visits, separated by 3 months
Population: Participants were censored if they started weight-altering medications, including glucagon-like peptide-1 receptor agonists, metformin, or insulin (n=4). Due to sample processing errors, n=2 additional results were missing.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Once Daily Text Message | Twice Daily Text Message | Fixed Step Count Goal | Ramped Step Count Goal | Loss Framed Incentive | Gain Framed Incentive | Daily Step Count Goal | Weekly Step Count Goal
Number analyzed (Participants) | 26 | 23 | 24 | 25 | 24 | 25 | 25 | 24
mg/dL | 0.0008 [-1.0 to 1.0] | 0.002 [-3.2 to 3.2] | 0.002 [-2.1 to 2.1] | 0.001 [-1.6 to 1.6] | 0.0005 [-0.5 to 0.5] | 0.004 [-3.9 to 3.9] | 0.002 [-1.7 to 1.7] | 0.001 [-1.2 to 1.2]
Statistical Analysis 1: Comparison: Once Daily Text Message vs Twice Daily Text Message; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-3.1 to 3.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fixed Step Count Goal vs Ramped Step Count Goal; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.0003, 95% CI 2-sided [-2.3 to 2.3] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Loss Framed Incentive vs Gain Framed Incentive; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-3.4 to 3.4] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Daily Step Count Goal vs Weekly Step Count Goal; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.0005, 95% CI 2-sided [-0.5 to 0.5] — [estimate comment as in outcome 1, analysis 4]

10. Secondary Outcome: Change in ALT
Description: U/L
Time Frame: From baseline to follow-up in-person study visits, separated by 3 months
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Once Daily Text Message | Twice Daily Text Message | Fixed Step Count Goal | Ramped Step Count Goal | Loss Framed Incentive | Gain Framed Incentive | Daily Step Count Goal | Weekly Step Count Goal
Number analyzed (Participants) | 25 | 24 | 24 | 25 | 24 | 25 | 24 | 25
U/L | 0.000000004 [-0.000008 to 0.000008] | 0.00000002 [-0.00003 to 0.00003] | 0.00002 [-0.03 to 0.03] | 0 [0 to 0] | 0 [0 to 0] | 0.00002 [-0.03 to 0.03] | 0.000003 [-0.004 to 0.004] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Once Daily Text Message vs Twice Daily Text Message; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = 0.00000001, 95% CI 2-sided [-0.00002 to 0.00002] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fixed Step Count Goal vs Ramped Step Count Goal; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.00002, 95% CI 2-sided [-0.03 to 0.03] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Loss Framed Incentive vs Gain Framed Incentive; Test type: Superiority — Main effects were estimated using generalized linear models with log link. No interactions were included (failure to converge).); Mean Difference (Final Values) = 0.00002, 95% CI 2-sided [-0.03 to 0.03] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Daily Step Count Goal vs Weekly Step Count Goal; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -0.000003, 95% CI 2-sided [-0.004 to 0.004] — [estimate comment as in outcome 1, analysis 4]

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 3 months
Description: Adverse events were assessed at study visits using questionnaires.
Arm/Group | 1FLD | 1FLW | 1RLD | 1RLW | 1FGD | 1FGW | 1RGD | 1RGW | 2FLD | 2FLW | 2RLD | 2RLW | 2FGD | 2FGW | 2RGD | 2RGW
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/4 | 0/5 | 0/4 | 0/3 | 0/3 | 0/4 | 0/4 | 0/5 | 0/5 | 0/4 | 0/4 | 0/4 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4 | 0/5 | 0/4 | 0/3 | 0/3 | 0/4 | 0/4 | 0/5 | 0/5 | 0/4 | 0/4 | 0/4 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 2/5 | 1/4 | 2/4 | 1/5 | 0/4 | 2/3 | 1/3 | 2/4 | 2/4 | 1/5 | 1/5 | 2/4 | 0/4 | 2/4 | 0/5 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1FLD (N=5) | 1FLW (N=4) | 1RLD (N=4) | 1RLW (N=5) | 1FGD (N=4) | 1FGW (N=3) | 1RGD (N=3) | 1RGW (N=4) | 2FLD (N=4) | 2FLW (N=5) | 2RLD (N=5) | 2RLW (N=4) | 2FGD (N=4) | 2FGW (N=4) | 2RGD (N=5) | 2RGW (N=4)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participant reported new diagnosis of anemia
Hypobetalipoproteinemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant was diagnosed with hypobetalipoproteinemia
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participants reported injuries related to minor trauma
stress fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant reported stress fracture in foot
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participant reported asthma exacerbation not requiring hospitalization
Skin irritation or rash on wrist (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participants reported minor skin irritation or rash associated with Fitbit wear on wrist
Skin irritation or rash, unspecified (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Generalized rash
Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participants reported mild viral or bacterial illnesses, not requiring hospitalization
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participant reported a migraine that required medical evaluation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT04874415/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT04874415/ICF_000.pdf